CLINICAL TRIAL: NCT07062302
Title: A Preliminary Efficacy Study on the Effectiveness of Low-Level Light Therapy for Vocal Fatigue
Brief Title: Effectiveness of Low-Level Light Therapy for Vocal Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Law, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC2023.483
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Vocal Fatigue
Keywords: vocal fatigue; voice disorders; photobiomodulation; low-level light therapy
MeSH Terms: conditions — Voice Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Photobiomodulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photobiomodulation arm (Experimental)
  Interventions: Device: photobiomodulation

INTERVENTIONS:
Device: photobiomodulation — The output of the photobiomodulation device is listed as below:
  * Irradiation size: 15 cm × 10 cm
  * Dual-wavelength: 660 nm + 850 nm
  * Optical power density: 10 - 15 mW/cm2
  * Dose density: 6J/cm2
  Other Names: low level light therapy

SUMMARY:
The goal of this phase 2 clinical trial is to examine the effectiveness of photobiomodulation in patients with vocal fatigue.

The main question it aims to answer is whether photobiomodulation is able to alleviate vocal fatigue in patients with diagnosed vocal fatigue.

Participants will ask to receive photobiomodulation treatment for 12 sessions over a three week period.

DETAILED DESCRIPTION:
Vocal fatigue is a common complaint of patients with voice disorder and is related to functional and/or organic voice disorders. Professional voice users, such as teachers and singers and actors, are particularly prone to vocal fatigue. It has been reported that vocal fatigue also associated with limitation to voice activities and participation. In patients with vocal fatigue, experience of inflammation and muscle pain are among possible symptoms and manifestations of the condition.

In literature, various definitions have been suggested for vocal fatigue. Welham and Maclagan defined vocal fatigue as the negative vocal adaptation led by prolonged use of voice, and it can consist of perceptual, acoustic or physiologic components of undesirable or unexpected functional changes in the laryngeal mechanism.

In exploring the nature of vocal fatigue, Titze capitalised on a generally recognised mechanism of muscle fatigue which comprised of a peripheral component and a central component. Specifically, for the peripheral component, fatigue may take place at the myo-neural junction, muscle membrane and endo-plasmic reticulum (i.e., the transmission mechanism) or the muscle filaments (i.e., the contractile mechanism), where depletion or accumulation of biochemical substances such as glycogen occurs.

Low-level light therapy (LLLT), also known as photobiomodulation (PBM) therapy, has been developed as a therapeutic procedure which involves the exposure to low levels of red and near infrared light to cells or tissues. It has been approved by the Food and Drug Administration (FDA) of the United States for aesthetic and medical purposes.

Ever since, it has been established as a non-invasive and safe approach for a number of medical processes, such as reducing inflammation, relieving pain, wound healing, skeletal muscle repair and treating neurological disorders. Specifically, its effectiveness on treating muscle fatigue was investigated with the focus placed on muscles such as bicep braquialis, quadriceps and orbicularis oris.

These studies utilised the feature of LLLT to interact with muscle tissues and therefore provide physiological and/or therapeutics effects to reduce muscle fatigue and enhance muscle performance. Relating this to the fatigue resulting from prolonged voice use at the laryngeal level, it is possible for LLLT to be developed as a treatment approach for vocal fatigue.

In a Phase 1 study, the potential effectiveness of using LLLT in vocal fatigue treatment by applying red or infrared Lights to healthy individuals following vocal loading tasks was explored. The authors concluded that red light might be effective in improving vocal fatigue on aspects of acoustic, aerodynamic, and self-perceptual markers.

The proposed study will be a Phase 2 behavioural study-controlled trial on the effectiveness of LLLT on treating vocal fatigue.

The primary objective of this study is to investigate the effectiveness of lower-level light therapy on reducing vocal fatigue on self-perceptual phenomena exhibited by participants, as well as acoustic and aerodynamic changes in voice.

Vocal Fatigue Index (Hong Kong-Chinese Version) (VFI(HK)) will be used as the primary outcome measurement methods. Perceptual evaluation of voice, acoustic measurement, aerodynamics evaluation (by maximum phonation time (MPT)), vocal symptoms scale and Voice Handicap Index (VHI-30) will be used as secondary outcome measurements.

The current study will be a preliminary clinical trial to identify the therapeutic efficacy of PBM on laryngeal muscles as a new treatment for patients with vocal fatigue. It could act as a pilot study and results obtained could be a foundation for Phase 3 RCT studies to investigate using LLLT to treat vocal fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old
* Meeting the diagnosis of vocal fatigue as per the VFI-HK
* Able to make informed consent
* Have not received any voice therapy before

Exclusion Criteria:

* History of photoallergy
* Significant medical or chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-03-09 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Vocal Fatigue Measure: Vocal Fatigue Index (VFI-HK) | This will be measured at baseline (pre-treatment) and within 2-weeks after the completion of treatment (post-treatment).
  The VFI(HK) contains 19 items in three domains (i) tiredness of voice and avoidance of voice use (ii) physical discomfort and (iii) improvement of symptoms after rest. All items are rated on a scale from zero (0, meaning "never") to four (4, meaning "always"). The score ranges from 0 to 76, with higher score indicating worst outcome.

SECONDARY OUTCOMES:
Vocal function measure: Voice Handicap Index - 30 | This will be measured at baseline (pre-treatment) and within 2-weeks after the completion of treatment (post-treatment).
  The VHI-30 contains 30 items in three subscales, namely "Functional", "Physical " and "Emotional". All items are rated on a scale from zero (0, meaning "never") to four (4, meaning "always"). The highest possible score for the VHI-30 is therefore 129, with the higher indicating worst scores.
Vocal Function Measure: Aerodynamic assessment | This will be measured at baseline (pre-treatment) and within 2-weeks after the completion of treatment (post-treatment).
  Maximum phonation time will be used as the aerodynamic measure. Maximum phonation will be measured in seconds (time), with the higher score indicated better outcome.
Vocal Function Measures: Acoustic voice analysis | This will be measured at baseline (pre-treatment) and within 2-weeks after the completion of treatment (post-treatment).
  Four parameters will be measures:
  (i) Jitter - Jitter represents the cycle-to-cycle variation in the fundamental frequency of the voice signal. Healthy, sustained phonation in young adults typically shows jitter values between 0.5% and 1.0%. Values above 1% may suggest dysphonia.
  (ii) Shimmer: Shimmer represents the cycle-to-cycle variation in the amplitude of the voice signal. Shimmer values below 3% are generally considered normal. Higher shimmer values can indicate dysphonia.
  (iii) Harmonic to noise ratio: HNR quantifies the ratio of harmonic to noise components in the voice signal. A high HNR indicates a strong presence of harmonics, which is characteristic of a clear, healthy voice. A low HNR suggests a greater proportion of noise in the voice, which is often associated with hoarseness.
  (iv) CPPS: CPPS measures the prominence of the cepstral peak, which represents the periodicity in the voice signal. Lower CPPS values suggest dysphonia.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the investigator, TL, upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2025

REFERENCES:
- [Background] Moreno M, Calvache C, Cantor-Cutiva LC. Systematic Review of Literature on Prevalence of Vocal Fatigue Among Teachers. J Voice. 2025 Jan;39(1):105-112. doi: 10.1016/j.jvoice.2022.07.029. Epub 2022 Sep 20. PMID 36137877
- [Background] Welham NV, Maclagan MA. Vocal fatigue: current knowledge and future directions. J Voice. 2003 Mar;17(1):21-30. doi: 10.1016/s0892-1997(03)00033-x. PMID 12705816